CLINICAL TRIAL: NCT04699227
Title: CAN REMOTE ISCHAEMIC CONDITIONING REDUCE INFLAMMATORY MARKERS IN COVID-19 PATIENTS - A MULTI-SITE, RANDOMISED PILOT STUDY
Brief Title: Can RIC Prevent Deterioration to Critical Care in Covid19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derek Yellon (Other)
Responsible Party: Sponsor-Investigator, Derek Yellon, Professor, University College London Hospitals
Organization: University College London Hospitals (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 20/SC/0192
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Covid19; Ischemia
Keywords: Covid19; Ischemia
MeSH Terms: conditions — COVID-19; Ischemia | interventions — Inflation, Economic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group not receiving RIC (Sham Comparator): Those randomised to the control group will have the blood pressure cuff placed on the arm, but it will not be inflated.
  Interventions: Other: Sham inflation
- Interventional group receiving RIC (Experimental): RIC will consist of 3-4 cycles of cuff inflations to 200 mmHg for 5 min with deflation to 0 mmHg for another 5 min, which is automatically administered by the pre-programmed cuff.
  Interventions: Procedure: Cuff application with inflation

INTERVENTIONS:
Procedure: Cuff application with inflation — The blood pressure cuff will be placed on the arm and inflated.
  Arms: Interventional group receiving RIC
Other: Sham inflation — The blood pressure cuff will be placed on the arm and not inflated.
  Arms: Control group not receiving RIC

SUMMARY:
The coronavirus disease (COVID-19) emerged in late 2019 and has since been diagnosed in over a million persons worldwide. As this virus progresses, it causes an extreme and uncontrolled response from the patient's immune system accompanied by reduced oxygen flow to major organs, and subsequent ischaemic injury.

The current treatment of COVID-19 is largely supportive without any cure or vaccine available at this time. Developing new methods to reduce this heightened inflammatory response is essential to halting progression of COVID-19 in patients and reducing the severity of damage.

The cellular mechanisms seen in COVID-19 are similar to those seen in patients with sepsis. A process known as Remote Ischemic Conditioning (RIC) is an intervention which has been shown to prevent cellular injury including those associated with sepsis. Based on the evidence from studies looking at sepsis, it is anticipated the same benefit would be seen in patients diagnosed with COVID-19.

RIC is a simple, non-invasive procedure where a blood pressure cuff is applied to the arm for repeated cycles of inflating and deflating (typically 3-5 cycles of 5 minutes each). This process activates pro-survival mechanisms in the body to protect vital organs and improve the immune system. Therefore, we believe it represents an exciting strategy to protect organs against reduced blood flow and extreme immune response, as seen in COVID-19 infections.

This study has already been fully approved

DETAILED DESCRIPTION:
COVID-19 has an early phase and a late, with rapid progression to ARDS (due to cytokine storm), multi-organ failure and death. Suppressing these cytokine elevations maybe a key to improved outcomes. Acute and Chronic (repeated) RIC has been shown to benefit in reducing the levels cytokines following LPS-induced sepsis in animal models (1). Furthermore, mortality was significantly reduced, following chronic RIC administration as opposed to acute RIC administration.

RIC in COVID-19 patients is a pilot, multi-centre, randomised study, designed to ascertain whether RIC decreases the severity of inflammatory markers associated with a "storm" score.

20 adult patients admitted to either The Royal Free or The Lister Hospital (Stevenage) with diagnosed COVID-19 will be enrolled into the study, of confirmed but not critical status. After enrolment, patients will be randomised (n = 10 per group) 1:1 to receive RIC or no adjunctive intervention.

RIC will consist of 3-4 cycles of cuff inflations to 200 mmHg for 5 min with deflation to 0 mmHg for another 5 min, which is automatically administered by the pre-programmed cuff. Those randomised to the control group will have the blood pressure cuff placed on the arm, but it will not be inflated. RIC will be performed daily for 15 days.

Venous blood will be collected following RIC administration (where possible) and saved for the subsequent measurement of inflammatory markers such as TNF, IL-1β, IL-6, and HMGB1 in addition to cardiac biomarkers Troponin T and NT pro terminal BNP. All biomarker analysis will occur at The Hatter Cardiovascular Institute, UCL.

The endpoint is area under the curve of inflammatory markers and cardiac biomarkers. Secondary endpoint will be the need for intensive care admission or death.

It would be our intention to use autoRIC devices (CellAegis, Canada) to ascertain whether RIC can lower the cytokine response. These devices are specifically designed, blood-pressure cuffs pre-programmed for the number of uses required by each patient; the intent being "a single patient-multiple use" cuff.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients (aged 18 - 80 yrs) with diagnosed COVID-19.

Exclusion Criteria:

* Contraindication for the use of a brachial cuff on either arm.
* Intercurrent disease with an expected life expectancy of less than 24 h, cardiac arrest, - Pregnant or breastfeeding women.
* Bleeding disorder or platelet count below 50.
* Currently enrolled in another research study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | 12 months
  The primary outcome is to demonstrate that remote ischaemic conditioning reduces the severity of inflammatory cytokine release which are responsible for the cytokine "storm" that occurs in following COVID-19 infection.
  The endpoint is area under the curve of inflammatory markers and cardiac biomarkers.

SECONDARY OUTCOMES:
Secondary Endpoint | 12 months
  Secondary endpoint will be the need for intensive care admission or death.

CONTACTS AND LOCATIONS:
Locations (4):
- Atherosclerosis and Vascular Biology laboratory, State University of Campinas, Campinas, Brazil
- Groote Schuur Hospital and Faculty of Health Sciences, University of Cape Town, Cape Town, South Africa
- United Kingdom (2):
  - Royal Free London NHS Foundation Trust,, London
  - East and North Hertfordshire NHS TrusEast and North Hertfordshire NHS Trus, Stevenage

IPD SHARING:
Plan to Share IPD: No
No identifiable, personal data will be collected as part of this study.

REFERENCES:
- [Derived] Lukhna K, do Carmo HRP, Castillo AR, Davidson SM, Geffen H, Giesz S, Golforoush P, Bovi TG, Gorag D, Salama A, Imamdin A, Kalkhoran S, Lecour S, Perroud MW Jr, Ntsekhe M, Sposito AC, Yellon DM. Effect of Remote Ischaemic Conditioning on the Inflammatory Cytokine Cascade of COVID-19 (RIC in COVID-19): a Randomized Controlled Trial. Cardiovasc Drugs Ther. 2024 Jun;38(3):433-445. doi: 10.1007/s10557-022-07411-2. Epub 2022 Nov 29. PMID 36445625
- [Derived] Davidson SM, Lukhna K, Gorog DA, Salama AD, Castillo AR, Giesz S, Golforoush P, Kalkhoran SB, Lecour S, Imamdin A, do Carmo HRP, Bovi TG, Perroud MW Jr, Ntsekhe M, Sposito AC, Yellon DM. RIC in COVID-19-a Clinical Trial to Investigate Whether Remote Ischemic Conditioning (RIC) Can Prevent Deterioration to Critical Care in Patients with COVID-19. Cardiovasc Drugs Ther. 2022 Oct;36(5):925-930. doi: 10.1007/s10557-021-07221-y. Epub 2021 Jun 25. PMID 34169381